CLINICAL TRIAL: NCT04448015
Title: Perinatal Care and Medication Assisted Treatment: Carbon/Emery Counties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jerry Cochran, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: A02769
Record Dates: First submitted 2020-06-18; First posted 2020-06-25 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Opioid-use Disorder; Pregnancy Related
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Perinatal Care (Experimental): Pregnant women enrolled in the study will receive enhanced perinatal care from community healthcare providers that have participated in the perinatal OUD education curriculum.
  Interventions: Other: Perinatal Opioid Use Disorder Education and Enhanced Perinatal Care

INTERVENTIONS:
Other: Perinatal Opioid Use Disorder Education and Enhanced Perinatal Care — University of Utah clinicians will provide face-to-face, online, and written training materials for health, mental health, and substance use service providers in Carbon and Emery Counties, UT.

SUMMARY:
The purpose of this study is to enhance perinatal opioid use disorder (OUD) treatment in a rural setting by developing an evaluated curriculum of perinatal OUD provider education.

DETAILED DESCRIPTION:
The research team will establish and evaluate a perinatal model of care for OUD serving two counties, Carbon and Emery, which have high rates of OUD and overdose. This model of care will entail University of Utah medical clinicians providing education and webinars to healthcare providers in Carbon/Emery counties who care for pregnant women with OUD and their babies. This model of care will also help other social and behavioral health care providers in the area to understand how to treat and better coordinate care. No clinical services are being provided by University of Utah investigators or staff.

ELIGIBILITY:
Provider Inclusion Criteria:

* Must be employed as staff at one of our sub-contracted agencies or community partners
* Must directly provide care to pregnant women with OUD in Carbon and/or Emery Counties, UT

Provider Exclusion Criteria:

* Unwilling or unable to adopt treatment approaches presented from University of Utah clinicians to patient care
* Not directly working with pregnant patients with OUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Self-report of linkage and adherence to treatment as assessed by the Treatment Service Review- 6 (TSR-6) | This data will be collected from each participant during a baseline assessment, a pre-delivery assessment occurring between 34 and 40 weeks of gestation, and a final assessment conducted within 30-days following delivery.
  Patients will complete the Treatment Services Review-6 (TSR-6) in order to measure changes in service across time. The TSR-6 is a clinically validated 56-item measure with excellent reliability for assessing drug and alcohol treatment engagement, medication use (including drug, alcohol, psychiatric, and physical health medications), psychiatric care, family services, financial/employment/housing, and legal services. This measure captures linkage/retention in care, that is to say: initiation and daily engagement in services. Specifically, the research team will capture frequency of meetings/sessions/days in OUD and other substance counseling and psychiatric care and social services. The research team will also use the TSR-6 medication use section to capture adherence to buprenorphine or methadone. Data collected will be used to measure change across time in linkage and retention in health and behavioral health services.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Utah Women's Health LLC, Price, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bryan MA, Smid MC, Cheng M, Fortenberry KT, Kenney A, Muniyappa B, Pendergrass D, Gordon AJ, Cochran G. Addressing opioid use disorder among rural pregnant and postpartum women: a study protocol. Addict Sci Clin Pract. 2020 Oct 31;15(1):33. doi: 10.1186/s13722-020-00206-6. PMID 33129355